CLINICAL TRIAL: NCT05793749
Title: Early Intervention to Prevent Gynecological Malignant Tumors Clinical Study of Lymphedema of the Lower Limbs in Patients With Radiotherapy After Lymphadenectomy
Brief Title: Early Intervention to Prevent Lower Limb Lymphedema of Gynecological Malignancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, professor，Doctor, Chongqing University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CQGOG0108
Record Dates: First submitted 2022-07-29; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Uterine Cervical Neoplasms; Endometrial Neoplasms; Lymphedema; Treatment Effectiveness
Keywords: Lymphedema; Endometrial Neoplasms; Uterine Cervical Neoplasms; Treatment Effectiveness
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Lymphedema

STUDY DESIGN:
Intervention Model Description: Random grouping (A:B=3:1): A: intervention group; B: nonintervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic lymphedema treatment (Experimental): Prophylactic lymphedema treatment：The lymphedema prophylaxis treatment consists of four parts:manual lymphatic drainage, skin care, functional exercise, and wearing lymphedema preventive compression stockings.
  The prophylactic lymphedema treatment group receives lymphedema prophylaxis twice a week for a total of 10 sessions, each requiring an interval of at least 48 hours but no more than 2 weeks.
  Interventions: Behavioral: Prophylactic lymphedema treatment
- Standard of care (No Intervention): Standard of care，includeIn knowledge education and telephone follow-up were routinely conducted.

INTERVENTIONS:
Behavioral: Prophylactic lymphedema treatment — 1. perform manual lymphatic drainage twice a week after the start of radiotherapy for a total of 10 times, and wear lymphedema compression stockings after each manual lymphatic drainage, 2. teach patients how to care for their skin. 3. perform functional exercises for lymphedema of the lower extremities twice a day for 15 ~ 20 minutes each time. 4. follow up observation: before the start of radiotherapy, every Friday during radiotherapy, and every 3 months after the end of radiotherapy, the occurrence of lymphedema and related symptoms and quality of life were evaluated.
  Arms: Prophylactic lymphedema treatment

SUMMARY:
This study is a prospective, randomized, controlled clinical trial of a single center in China and plans to enroll 400 patients.

1. Patients with diagnosed gynecological malignancies who underwent pelvic and abdominal lymphadenectomy and required pelvic radiotherapy;
2. Random grouping (A:B=3:1): A. Prophylactic lymphoedema treatment; B. Standard care group;
3. Preventive lymphedema health education was given to patients with gynecological malignant tumors without contraindications before surgery. All patients were randomly divided into an intervention group and a nonintervention group. The intervention group received preventive lymphedema treatment twice a week. 10 times, and the interval between the two treatments was not less than 48 hours and not more than 2 weeks. The intervention measures included four parts: manual lymphatic drainage, skin care, functional exercise, and wearing lymphedema preventive compression stockings. In the nonintervention group, knowledge education and telephone follow-up were routinely conducted.
4. All patients were evaluated for edema, lymphedema symptoms and quality of life 1 day before radiotherapy, every Friday during radiotherapy and every 3 months thereafter. Bioelectrical impedance measurement and leg diameter measurement were used to evaluate edema, the Gynecologic Cancer Lymphedema Questionnaire (GCLQ) was used to evaluate lymphedema symptoms, and the EORTC Quality of Life Scale (QLQ-C30) was used to evaluate quality of life. followed up to 2 years after the end of lymphedema prophylaxis.

DETAILED DESCRIPTION:
Research background Gynecological malignancies, including cervical cancer, ovarian cancer, endometrial cancer, vulvar cancer, etc., are important diseases threatening women's health worldwide, and their main treatment methods are surgery and radiotherapy. During surgery, different numbers of lymph nodes are removed, and lymphatic fluid and tissue exudate from the stump lymphatic vessels accumulate, causing disruption of the original lymphatic circulation and obstruction of lymphatic fluid return, which leads to lower limb edema . The longer the radiotherapy lasts, the more serious the phenomenon of collateral circulation will be, and the lymphatic return pathway will be damaged, resulting in lower limb lymphedema .

Lower extremity lymphedema is a relatively common complication after treatment for gynecologic malignancies, and it has been reported that approximately 20 million patients worldwide are affected by lower extremity lymphedema. The overall incidence of lower extremity lymphedema after gynecologic malignancy treatment is about 25% and can be as high as 70% in special groups . Age, weight, radiotherapy dose, duration of postoperative radiotherapy, tumor stage, daily standing time, number of lymph node dissection, and co-infection are all risk factors for the occurrence of lower extremity lymphedema.

Lymphedema is characterized by sunken edema at the beginning of the disease and progresses to include swelling, numbness, heaviness, tissue fibrosis, impaired movement, and rough epidermal keratinization, and increases the risk of inflammation of the lymphatic vessels and surrounding tissues and cellulitis. Lower extremity lymphedema is a chronic progressive disease that is difficult to cure and has a negative impact on limb function, daily life, quality of life and psychological well-being.

The treatment of lymphedema includes surgical treatment and conservative treatment. The conservative treatment methods include Complex Decongestion Therapy (CDT), external application of Chinese herbal medicine and western medicine, etc. The Complex Decongestion Therapy (CDT) is the most widely used lymphedema treatment with the best efficacy internationally in recent years. The treatment method, but requires long-term or even lifelong care , which brings huge psychological burden and economic pressure to the patient's family. Therefore, lymphedema of the lower extremities should be prevented, and preventive and therapeutic measures should be taken as early as possible to improve the quality of life of patients.

Currently, studies on lymphedema prevention have focused on interventions for breast cancer-related lymphedema , while few studies have been reported on the prevention of lymphedema associated with gynecologic malignancies. Research reported that early intervention with freehand lymphatic drainage technique could effectively prevent lower limb lymphedema, and Research showed that full range of hip exercises could prevent lower limb lymphedema after cervical cancer surgery, in addition, some studies also found that freehand lymphatic drainage combined with Kegel training could prevent vulvar stage I lymphedema after cervical cancer surgery, however, these studies have some limitations, such as small sample size and limited study content. However, these studies have limitations, such as small sample size and limited study content. Moreover, there are no empirical studies on the prevention of lower extremity lymphedema in large samples, and there is no unified standard for the prevention and management of lower extremity lymphedema. Therefore, in this study, the investigators used an evidence-based approach and clinical experience to conduct a prospective study on the prevention of lower limb lymphedema in order to reduce the incidence of lower limb lymphedema, improve patients' quality of life, and reduce their economic burden.

Research objective

1. To understand the incidence of lymphedema after gynecological tumor surgery and radiotherapy and its impact on the quality of life of patients.
2. Through preventive lymphedema treatment intervention, reduce the proportion of lymphedema, reduce the economic burden of patients, and improve their quality of life.
3. We aimed to find a more economical and effective method to treat gynecological malignant tumor lymphedema.

Main outcome measures: The incidence of lower extremity lymphedema after gynecological cancer surgery and radiotherapy, and the incidence of lower extremity lymphedema after prophylactic lymphedema treatment.

Secondary outcome measures: quality of life, incidence of lymphedema symptoms, and progression-free survival (PFS).

Study population

Inclusion criteria:

1. Gynecologic oncology patients undergoing radiotherapy after lymph node surgery who voluntarily participate in this study and sign an informed consent form.
2. 18 to 60 years old.
3. Eastern Cooperative Oncology Group（ECOG) score less than 2.
4. Expected survival time greater than 3 years.
5. Hemoglobin(Hb) greater than or equal to 70 g/L, white blood cells (WBC)greater than or equal to 3.5 × 109 /L, neutrophils(ANC)greater than or equal to 1.5 × 109 /L, platelets (PLT)greater than or equal to 80 × 109 /L.
6. serum alamine aminotransferase(ALT) and glutamic oxalacetic transaminase(AST) less than 2 times the normal value and creatinine less than 1.5 times the normal value, albumin greater than or equal to 35g/L.
7. Women of childbearing potential must have had a pregnancy test (serum or urine) within 7 days prior to enrollment and have a negative result and be willing to use an appropriate method of contraception for the duration of the trial.
8. Ability to comply with the trial protocol, as judged by the investigator.

Exclusion criteria:

1. Lymphedema and deep vein thrombosis of the lower extremities were clearly diagnosed;
2. Acute infection of any kind;
3. Patients with lower extremity edema;
4. pregnancy, menstrual period;
5. Recent major abdominal surgery (determined by the investigator);
6. Radiation colitis, cystitis, intestinal infection, small bowel or large bowel diverticulitis or diverticulitis;
7. Liver fibrosis;
8. Abdominal aortic aneurysm;
9. acute phlebitis;
10. Severe arterial obstructive disease, arterial ulcer, ABPI (ankle-brachial blood pressure index) greater than 1.3 and less than 0.5;
11. Severe peripheral neuropathy;
12. Poor control of hypertension, poor control of stroke and diabetes, and severe bronchial asthma;
13. Patients who cannot understand the experimental content and cannot cooperate and those who refuse to sign the informed consent;
14. Those with concomitant diseases or other special circumstances that seriously endanger the patient's safety or affect the patient's completion of the study.

Subject Termination Criteria

1. The investigator believes that the treatment should be terminated from the perspective of the best benefit of the patients;
2. There are intolerable adverse reactions, after confirmation by the investigator;
3. Failure to complete the treatment according to the cycle and time;
4. The patient withdraws informed consent.

Elimination criteria:

(1) Those who did not meet the standards and were mistakenly included.

ELIGIBILITY:
Inclusion Criteria:

1.Gynecologic oncology patients undergoing radiotherapy after lymph node surgery who voluntarily participate in this study and sign an informed consent form.

2.18 to 60 years old. 3.Eastern Cooperative Oncology Group（ECOG) score less than 2. 4.Expected survival time greater than 3 years. 5.Hemoglobin(Hb) greater than or equal to 70 g/L, white blood cells (WBC)greater than or equal to 3.5 × 109 /L, neutrophils(ANC)greater than or equal to 1.5 × 109 /L, platelets (PLT)greater than or equal to 80 × 109 /L.

6.serum alamine aminotransferase(ALT) and glutamic oxalacetic transaminase(AST) less than 2 times the normal value and creatinine less than 1.5 times the normal value, albumin greater than or equal to 35g/L.

7.Women of childbearing potential must have had a pregnancy test (serum or urine) within 7 days prior to enrollment and have a negative result and be willing to use an appropriate method of contraception for the duration of the trial.

8.Ability to comply with the trial protocol, as judged by the investigator.

Exclusion Criteria:

1. Lymphedema and deep vein thrombosis of the lower extremities were clearly diagnosed;
2. Acute infection of any kind;
3. Patients with lower extremity edema;
4. pregnancy, menstrual period;
5. Recent major abdominal surgery (determined by the investigator);
6. Radiation colitis, cystitis, intestinal infection, small bowel or large bowel diverticulitis or diverticulitis;
7. Liver fibrosis;
8. Abdominal aortic aneurysm;
9. acute phlebitis;
10. Severe arterial obstructive disease, arterial ulcer, ABPI (ankle-brachial blood pressure index) greater than 1.3 and less than 0.5;
11. Severe peripheral neuropathy;
12. Poor control of hypertension, poor control of stroke and diabetes, and severe bronchial asthma;
13. Patients who cannot understand the experimental content and cannot cooperate and those who refuse to sign the informed consent;
14. Those with concomitant diseases or other special circumstances that seriously endanger the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The indication was for patients with gynecological malignancy
Enrollment: 400 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2026-07-29 (Estimated); Study Completion 2026-07-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of lymphedema | Incidence of lymphedema in the prophylactic lymphedema treatment group and the standard treatment group at 2 years after the end of radiotherapy
  The incidence of lower extremity lymphedema after gynecological cancer surgery and radiotherapy, and the incidence of lower extremity lymphedema after prophylactic lymphedema treatment.
Quality of life of patients | Quality of life QLQ-C30 scores for the prophylactic lymphedema treatment group and the standard treatment group at 2 years after the end of radiotherapy
  The quality of life of cancer patients (QLQ-C30) was used to assess the quality of life of patients. Including the overall quality of life subscale, functional subscale, symptom subscale, and individual test items. The higher the overall quality of life subscale and the functional subscale score, the better the quality or function. The more severe the symptoms.

SECONDARY OUTCOMES:
Subjective feelings | Quality of life GCLQ scores for the prophylactic lymphedema treatment group and the standard treatment group at 2 years after the end of radiotherapy
  The Gynecologic Cancer Lymphedema Questionnaire (GCLQ) was used to evaluate the subjective feelings of patients, which was mainly used to evaluate whether the limbs had symptoms such as swelling, pain, and heaviness. The evaluation included 7 symptom groups of heaviness, edema (overall), swelling (local), infection-related symptoms, pain, numbness, and limb function, with a total of 20 items.1 mark for "yes" and 0 mark for "no" for each entry. The higher the GCLQ score, the worse the subjective perception, and a score greater than or equal to 4 is recognized as the onset of lymphedema.
2-year progression-free survival,2-year PFS | 2-year PFS was defined as the time from randomization to the first occurrence of disease progression or death from any cause within 2 years
  2-year PFS was defined as the time from randomization to the first occurrence of disease progression or death from any cause within 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
This study is a prospective, randomized, controlled clinical trial of a single center in China and plans to enroll 400 patients. 1.Patients with diagnosed gynecological malignancies who underwent pelvic and abdominal lymphadenectomy and required pelvic radiotherapy. 2.Random grouping (A:B=3:1).
  3.Preventive lymphedema health education was given to patients with gynecological malignant tumors without contraindications before surgery. 4.All patients were evaluated for edema, lymphedema symptoms and quality of life ,Bioelectrical impedance measurement and leg diameter measurement , the Gynecologic Cancer Lymphedema Questionnaire (GCLQ) , and the EORTC Quality of Life Scale (QLQ-C30) will be used

REFERENCES:
- [Result] Cortez AJ, Tudrej P, Kujawa KA, Lisowska KM. Advances in ovarian cancer therapy. Cancer Chemother Pharmacol. 2018 Jan;81(1):17-38. doi: 10.1007/s00280-017-3501-8. Epub 2017 Dec 16. PMID 29249039
- [Result] Minion LE, Tewari KS. Cervical cancer - State of the science: From angiogenesis blockade to checkpoint inhibition. Gynecol Oncol. 2018 Mar;148(3):609-621. doi: 10.1016/j.ygyno.2018.01.009. Epub 2018 Feb 3. PMID 29666026
- [Result] 李可心，孙洪赞，辛军，等.早期宫颈癌盆腔淋巴结转移危险因素及PET/CT诊断[J].中国医学影像技术，2018，34: 265-269.
- [Result] 朱认真，张开宇，李倩.宫颈癌术后放疗致下肢淋巴水肿及神经电生理功能的影响及机制分析[J]. 实用癌症杂志, 2020，35: 121-124
- [Result] Dessources K, Aviki E, Leitao MM Jr. Lower extremity lymphedema in patients with gynecologic malignancies. Int J Gynecol Cancer. 2020 Feb;30(2):252-260. doi: 10.1136/ijgc-2019-001032. Epub 2020 Jan 7. PMID 31915136
- [Result] Jiang X, Nicolls MR, Tian W, Rockson SG. Lymphatic Dysfunction, Leukotrienes, and Lymphedema. Annu Rev Physiol. 2018 Feb 10;80:49-70. doi: 10.1146/annurev-physiol-022516-034008. Epub 2017 Oct 13. PMID 29029593
- [Result] 张赫,孔为民.宫颈癌治疗后下肢淋巴水肿预防进展[J].国际妇产科学杂志,2021,48(02):139-143.
- [Result] Fukushima T, Tsuji T, Sano Y, Miyata C, Kamisako M, Hohri H, Yoshimura C, Asakura M, Okitsu T, Muraoka K, Liu M. Immediate effects of active exercise with compression therapy on lower-limb lymphedema. Support Care Cancer. 2017 Aug;25(8):2603-2610. doi: 10.1007/s00520-017-3671-2. Epub 2017 Apr 6. PMID 28386788
- [Result] 中华整形外科学分会淋巴水肿学组.外周淋巴水肿诊疗的中国专家共识[J].中华整形外科杂志,2020,36(4):355-360.
- [Result] 梁笑媚,黄伟斌.腋窝反向淋巴作图预防乳腺癌术后上肢水肿的预防应用研究[J].中国卫生标准管理,2021.12(15):58-60.
- [Result] 白巧玲,王星.宫颈癌术后早期徒手淋巴引流预防术后下肢淋巴水肿[J].现代肿瘤医学,2021,29(19):3440-3442.
- [Result] Carter J, Raviv L, Appollo K, Baser RE, Iasonos A, Barakat RR. A pilot study using the Gynecologic Cancer Lymphedema Questionnaire (GCLQ) as a clinical care tool to identify lower extremity lymphedema in gynecologic cancer survivors. Gynecol Oncol. 2010 May;117(2):317-23. doi: 10.1016/j.ygyno.2010.01.022. Epub 2010 Feb 16. PMID 20163847
- [Result] Taarnhoj GA, Kennedy FR, Absolom KL, Baeksted C, Vogelius IR, Johansen C, Velikova G, Pappot H. Comparison of EORTC QLQ-C30 and PRO-CTCAE Questionnaires on Six Symptom Items. J Pain Symptom Manage. 2018 Sep;56(3):421-429. doi: 10.1016/j.jpainsymman.2018.05.017. Epub 2018 May 25. PMID 29807157